CLINICAL TRIAL: NCT00919360
Title: Expression of Vascular Endothelial Growth Factor and Its Effectors in Preeclampsia
Brief Title: Gene Expression In Pregnancies Complicated by Preeclampsia
Status: Terminated | Type: Observational
Why Stopped: PI is no longer at University of Rochester, has moved to University of Florida, Gainesville. PI email now homonq@ufl.edu. Phone is 352-273-7675
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Monique Ho, Assistant Professor, University of Florida
Other Study IDs: RSRB# 22086
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, placental and decidual tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Gravidas without history of hypertension of any kind, and matched to cases for parity, gestational age, labor status, mode of delivery, maternal age, and race.
  Interventions: Procedure: collection of maternal blood specimen prior to delivery; Procedure: collection of placental cord blood after delivery; Procedure: collection of placental tissue; Procedure: collection of strip of decidua from uterine lining from cesarean section deliveries
- Preeclamptics: Gravidas at 32-42 weeks gestation, delivered by Caesarean Section, who have preeclampsia as defined by Sibai et al, 1997.
  Interventions: Procedure: collection of maternal blood specimen prior to delivery; Procedure: collection of placental cord blood after delivery; Procedure: collection of placental tissue; Procedure: collection of strip of decidua from uterine lining from cesarean section deliveries

INTERVENTIONS:
Procedure: collection of maternal blood specimen prior to delivery — approximately 5 cc. of maternal blood will be drawn prior to delivery
Procedure: collection of placental cord blood after delivery — approximately 5 cc. of fetal cord blood from the umbilical cord blood vessel will be collected after cord is clamped
Procedure: collection of placental tissue — within 10 minutes of delivery, the placenta will be radially transected, and a full-thickness slice from the central region removed using sterile technique by scalpel.This will be placed into a pre-prepared container of RNA preservation medium.
Procedure: collection of strip of decidua from uterine lining from cesarean section deliveries — A strip of decidua will be removed from the upper lip of uterine incision by the surgeon and placed in RNA preservation medium.

SUMMARY:
The purpose of this study is to figure out some of the differences in bodily function between women who have preeclampsia and those who do not.

* This may eventually lead to an understanding of its cause. At this time, there is no known way to prevent preeclampsia, and the cause is not known.
* The only treatment is delivery of the baby, even if it is premature, in order to decrease the risk to the mother.

DETAILED DESCRIPTION:
* Preeclampsia is a pregnancy-related disorder that occurs in about 6% of all pregnancies.
* In its mild for, preeclampsia involves high blood pressure. More severe forms of preeclampsia can lead to more serious pregnancy complications.
* At this time, there is no known way to prevent preeclampsia, and the cause is not known. The only treatment is delivery of the baby, even if it is premature, in order to decrease the risk to the mother.
* The purpose of this study is to figure out some of the differences in bodily function between women who have preeclampsia and those who do not. This may eventually lead to an understanding of its cause.

ELIGIBILITY:
Inclusion Criteria:

* Gravidas at 32-42 weeks gestation,who have preeclampsia as defined by Sibai et al, 1997.
* Control patients: Gravidas without history of hypertension of any kind, and matched to cases for parity, gestational age, labor status, maternal age, and race.

Exclusion Criteria:

* Prior betamethasone administration, fetal growth restriction (<3%ile), prior chronic hypertension (nonpregnant or < 20 weeks gestation any pregnancy), chorioamnionitis, major fetal anomaly or chromosome abnormality, multiple gestation, and maternal diabetes (any class except diet-controlled gestational).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gravidas at 32-42 weeks gestation who present to Labor and Delivery units at University of Rochester, Strong Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2008-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Relative pattern of expression in cases and matched controls of a robust set of genes in the VEGF/sFLT mediated model for preeclampsia in the placenta and decidua | 1- 2 years

SECONDARY OUTCOMES:
From this expression pattern,determine the validity of 18s ribosomal subunit as an endogenous control in this tissue. | 1- 2 years
Using relative expression analysis in an embedded set of control subjects, determine whether common variables e.g. labor, parity independently influence expression of these genes of interest in the tissues studied | 1 - 2 years
Determine the population variance for each gene of interest | 1 - 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pressman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States